CLINICAL TRIAL: NCT05668351
Title: Phase II Trial Of Sparing The Urethra, Pudendal Artery And Rectum During Stereotactic Ablative Body Radiotherapy (SUPR-SABR) for Low and Intermediate Risk Prostate Cancer
Brief Title: Stereotactic Ablative Radiation Therapy for Prostate Cancer
Acronym: SUPR-SABR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Harriet Eldredge-Hindy, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUPR-SABR 103629
Record Dates: First submitted 2022-12-06; First posted 2022-12-29 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: stereotactic body radiation therapy; stereotactic ablative body radiotherapy; SBRT; SABR; pudendal artery
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Stereotactic Ablative Body Radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SUPR-SABR treatment (Experimental): The prescription dose of this study will be 40 Gy in 5 fractions assigned to PTV_4000 which permits sparing of the rectum, urethra and pudendal artery. There will be a secondary dose level of 36.25 Gy in 5 fractions. A minimum dose of 36.25 Gy will be given to the entire prostate PTV_3625. 36.25 Gy in five fractions is currently endorsed as a standard of care for localized prostate cancer by the National Comprehensive Cancer Network guidelines in prostate cancer. Escalating the therapeutic radiation dose above 36.25 Gy provides potential for improved biochemical control of prostate cancer and decrease in relapse free survival.
  Interventions: Radiation: SUPR-SABR treatment

INTERVENTIONS:
Radiation: SUPR-SABR treatment — SUPR-SABR prescription dose to the PTV_4000 will be 8 Gy per fraction for five fractions. The prescription dose to PTV_3625 will be a minimum of 7.25 Gy per fraction for five fractions. SABR will be delivered 2-3 times a week, every other day. There will be a minimum of 40 hours between fractions and maximum of 128 hours between fractions.

SUMMARY:
This single arm trial will investigate a novel way to plan and deliver SABR for prostate cancer. Prostate-directed SABR will be high-dose SABR (40 Gy in 5 fractions) with central sparing of the urethra and peripheral sparing of the rectum and pudendal arteries (SUPR-SABR). This study tests the hypothesis that genitourinary (GU) and gastrointestinal (GI) toxicity rates following SUPR-SABR are comparable to (or possibly lower than) historical GU and GI toxicity rates following standard SABR (stSABR) with 36.25 Gy in the treatment of low- and intermediate-risk prostate cancer.

DETAILED DESCRIPTION:
It is estimated that there will be 268,000 prostate cancer diagnoses and nearly 35,000 deaths due to prostate cancer in the United States in 2022 [1]. Most men diagnosed with prostate cancer present with localized or organ confined disease which is most commonly managed with active surveillance, prostatectomy, brachytherapy, and external beam radiotherapy (EBRT). Conventionally fractionated (1.8-2.0 Gy per fraction for nine weeks) EBRT is of historical and clinical importance in localized prostate cancer, however, moderately hypofractionated (≥2.5 Gy per fraction for four to six weeks) EBRT and SABR have also emerged as standards of care in appropriately selected patients.

The increased precision associated with image guided stereotactic techniques now permits safe delivery of large doses per fraction, also known as hypofractionation. SABR is a specific type of hypofractionated RT. Hallmarks of the SABR technique, also commonly known as stereotactic body radiotherapy (SBRT), include doses of at least 5 Gy per fraction, five or fewer fractions, motion management, noncoplanar beam or arc therapy, body immobilization, and ablative prescription doses.

There is growing interest in the use of SABR in men with low- and intermediate- risk prostate cancer due to their lower risk of extra prostatic disease including pelvic lymph node micrometastases and the low alpha/beta ratio of prostate cancer. Several series with follow up times exceeding five years have demonstrated excellent biochemical control for SABR approaching 95% for low risk and 80-90% for intermediate risk disease with low rates of clinically significant late GU and GI toxicity. Most published clinical experiences of SABR for prostate cancer have employed 35 to 36.25 Gy in 7- to 7.25 Gy fractions (i.e., standard SABR or stSABR). Importantly, it has never been established whether this represents the optimal dose level for SABR and, nationally, there is not only a single standard of care for SABR prescription dose and fractionation. What is more, contemporary literature with prostate SABR suggests a benefit with dose escalation, however, there is interest in avoiding a parallel increase in GU, GI, and sexual side effects of treatment.

The proposed trial concept would offer men with low- and intermediate-risk prostate cancer a dose-escalated SABR regimen (SUPR-SABR) of 40 Gy in 5 fractions with a safety profile already supported by medical literature and which is expectedly more efficacious than stSABR. This dose and fractionation is already being used in some radiation oncology practices. However, to further improve the therapeutic index of curative RT, the protocol will employ all available methods to spare the urethra, pudendal artery, and rectum (SUPR-SABR): foley catheter placement during planning, rectal spacer gel placement, endorectal balloon during planning and treatment, prostatic immobilization, strict contouring and dose constraints, and the most highly conformal photon planning available. This protocol will offer men a clinical study with highly important endpoints and lower anticipated treatment related morbidity. If the primary analysis demonstrates favorable healthcare related quality of life (HRQOL) with SUPR-SABR when compared to prospectively collected historic controls of stSABR, then this would serve as the basis for a randomized trial between SUPR-SABR and stSABR.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male patients aged 18 years and older
4. In good general health as evidenced by medical history to be a candidate for curative-intent prostate cancer treatment
5. Ability to receive pelvic radiotherapy and be willing to adhere to the SUPR-SABR regimen
6. Previously untreated prostate cancer (with cytotoxic chemotherapy, surgical or radiation therapy)
7. Localized adenocarcinoma of the prostate with the following features:

   1. cT1-T2c
   2. PSA<20

      * Patients receiving a 5-alpha reductase inhibitor must have a PSA <10
   3. Grade Group 1-3
8. Patient willing and able to complete the EPIC questionnaire at time of registration and 1-, 12-, and 24- months post treatment
9. Prostate volume <120 cc
10. History and physical including a digital rectal exam 90 days prior to registration
11. ECOG performance status 0-2
12. Be eligible and willing to undergo MRI prostate and pelvis as a component of RT planning
13. Bone and soft tissue imaging as clinically indicated (for unfavorable intermediate risk or symptomatic patients only) within 120 days prior to registration
14. IPSS score ≤20 at time of initial history and physical with treating radiation oncologist

Exclusion Criteria:

1. Female patients (due to lack of prostate gland)
2. Concurrent use of testosterone supplementation
3. Known homozygous for ATM pathogenic mutation
4. Prior pelvic RT
5. Treatment with another investigational drug for prostate cancer
6. Pre-existing conditions or overall health status which disqualifies the patient from curative-intent RT
7. Prior or concurrent invasive pelvic malignancy (except non-melanomatous skin cancer) or lymphomatous or hematogenous malignancy, unless disease free for a minimum of 5 years
8. Patients with distant metastases from prostate cancer
9. Patients with lymph node involvement by prostate cancer
10. Prior prostatectomy, cryotherapy, high-intensity focused ultrasound, pelvic irradiation overlapping with fields needed for prostate cancer treatment, prostate brachytherapy, or previous cytotoxic chemotherapy for prostate cancer
11. Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — diagnosis of prostate cancer
Enrollment: 36 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
12 month Expanded Prostate Cancer Index Composite (EPIC) genitourinary score | 12 months
  EPIC score at 12 months post intervention will be compared with pre-intervention scores. Score scale is 0 to 100 with lower scores indicating more severe symptoms.
12 month Expanded Prostate Cancer Index Composite (EPIC) gastrointestinal score | 12 months
  EPIC score at 12 months post intervention will be compared with pre-intervention scores. Score is 0 to 100 with lower scores indicating more severe symptoms.

SECONDARY OUTCOMES:
24 month Expanded Prostate Cancer Index Composite (EPIC) genitourinary score | 24 months
  EPIC score at 24 months post intervention will be compared with pre-intervention scores. Score is 0 to 100 with lower scores indicating more severe symptoms.
24 month Expanded Prostate Cancer Index Composite (EPIC) gastrointestinal score | 24 months
  EPIC score at 24 months post intervention will be compared with pre-intervention scores. Score is 0 to 100 with lower scores indicating more severe symptoms.
Incidence of Common Terminology Criteria for Adverse Events (CTCAE) version 5 grade 3 or higher adverse events from radiation therapy | 24 months
  CTCAE adverse events are on a scale of 0 to 5 with 5 indicating the most severe events.
1 month genitourinary toxicity as assessed by the International Prostate Symptom Score (IPSS) | 1 month
  The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms. IPSS scores at 1 month will be compared with baseline pretreatment IPSS scores.
12 and 24 month erectile function as assessed by the Sexual Health Inventory for Men (SHIM) score. | 24 months
  SHIM score is on a scale of 5-25 with lower scores indicating more severe symptoms of erectile dysfunction.
Biochemical failure rate at 24 months. | 24 months
  Biochemical failure will be reported as a percentage. biochemical failure is defined as prostate specific antigen nadir post treatment + 2 ng/mL.
To correlate changes in Sexual Health Inventory for Men (SHIM) score at 12 and 24 months with radiation dose to the pudendal artery (Gy) | 24 months
  SHIM score is 5 to 25 with lower scores indicating worse erectile function

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Eldredge-Hindy, MD, Principal Investigator — MUSC Department of Radiation Oncology
Locations (1):
- Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No